

General Template - Drug Clinical Trial **Version Date: November 2022** 

| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

Protocol Title: A RANDOMIZED, BALANCED, PHASE 1, MULTIPLE-DOSE, OPEN-LABEL, TWO-TREATMENT, TWO-PERIOD, TWO-SEQUENCE, CROSSOVER, BIOAVAILABILITY RELATIVE STUDY TO **INVESTIGATE** BRAIN/PLASMA PHARMACOKINETICS AND SAFETY OF AN ALOO1 ORAL CAPSULE COMPARED TO A MARKETED IMMEDIATE-RELEASE LITHIUM CARBONATE CAPSULE IN HEALTHY ADULT SUBJECTS

Principal Investigator: Ovidiu Andronesi MD, PhD

Site Principal Investigator:

Description of Subject Population: Healthy subjects between the ages of 18 and 64

#### About This Consent Form

IRB Protocol No: 2024P003031

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

If you decide to take part in this research study, you must sign this form to show that you fully understand the requirements of the study and are willing to participate. We will give you a signed copy of this form to keep.

## **Key Information**

We are asking you to be in a research study, consisting of a 28-days screening period, two treatment periods of 16 days each – separated by a 9 to 28 days washout period – and a 4-week follow-up period after the second treatment period. This form will tell you what you should expect if you agree to be in the study. You will find more information about the research study and visit schedule later in this form.

It is your decision whether or not to join the study. We are asking you to be in this study because you are in good health. We are conducting this clinical trial to assess the safety and dosage of a new lithium formulation that could be helpful for people with psychiatric or neurological disorders. If you agree, you will take daily doses of either the investigational study drug (AL001) or a marketed Lithium Carbonate drug for 14 days while staying overnight at the research center on the main campus of Massachusetts General Hospital. You will also undergo a series of blood

IRB Expiration Date: 3/5/2026 Consent Form Valid Date: 5/21/2025 IRB Submission: AME4




| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

draws and MRI scans over a 24-hour period. You will then be released from the research center to begin the washout period prior to returning for the second treatment period. When you return to the research center for the second treatment period, you will repeat the above process with the alternate drug. You will be in the study for approximately 4 and a half months if you decide to complete the entire study.

The main risks of being in the study are fatigue, frustration, and feelings of isolation due to study procedures and design.

You will be paid up to \$10,300 via a debit card for completing the entire research study. You will find more information about the payment amount for each visit and a compensation plan if you do not complete all study visits later in this form.

Prior to signing this informed consent (and anytime afterwards), you can ask the study staff or call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Ovidiu Andronesi, MD, PhD is the person in charge of this research study. You can call him at (617) 643-6864, M-F 9am-5pm. You can also call the Study Nurse at (617) 643-8464, M-F 9am-5pm, or Alison McManus, DNP at (617) 643-4848, 24/7, with questions about this research study.

If you have questions about the scheduling of appointments or study visits, call the Study Coordinator at (617) 724-6094.

If you want to speak with someone **not** directly involved in this research study, please contact the Mass General Brigham IRB. You can call them at (857) 282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure perceived to take part in, or to continue in the research study




| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

### **Detailed Information**

A description of this clinical trial is available on ClinicalTrials.gov Web site (<a href="http://www.ClinicalTrials.gov/study/NCT06921590">http://www.ClinicalTrials.gov/study/NCT06921590</a>), as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### Why is this research study being done?

We are doing this research study to find out if AL001, a new crystalized form of Lithium, has a better absorption and metabolic profile than commonly used marketed lithium salts. We will also be monitoring any side effects that may arise when taking AL001.

AL001 is not approved by the U.S. Food and Drug Administration (FDA). This means that AL001's use in this research study is considered "investigational" and it can currently only be used in research studies.

About 64 healthy volunteers and volunteers with Alzheimer's disease have taken part in a prior research study to assess a safe and tolerable dose of AL001. In addition, 28 healthy volunteers participated in an initial safety study. AL001 was shown to be well tolerated and safe in both healthy and Alzheimer's disease populations.

This research study will compare AL001 (five crystallized lithium capsules/dose) to a comparable dose of Lithium Carbonate (one capsule/dose) given by mouth 3 times per day for 14 days. Lithium Carbonate is commonly used to treat neuropsychiatric conditions. During one of the 16-day treatment periods of the study you will receive AL001 capsules. During the other 16-day treatment period you will receive one capsule of Lithium Carbonate. There is a 9-28 days washout period between the two treatments. The treatment you start the study on will be assigned randomly (like a toss of a coin), but you will know which of the two drug products you are receiving during each treatment period.

## Who will take part in this research?

We are asking you to take part in this research study because you are between the ages of 18 and 64 and are not suffering from any chronic or current medical conditions. This study will only involve healthy volunteers.

About 6 participants will take part in this research study. All participants will take part in this study at Massachusetts General Hospital (MGH).

Alzamend Neuro, Inc. is the sponsoring company paying for this research to be done.





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

#### How long will you take part in this research?

It will take you about 4 and a half months to complete this research study. This research study consists of an in-person screening period, two 16-day (overnight) treatment periods separated by a washout period, and a follow up period. The two treatment periods in the study will involve each a 16-day, 15-night (overnight) stay, mainly occurring at Massachusetts General Hospital's main campus within the Translational and Clinical Research Centers (TCRC). The last overnight stay for each treatment period will occur at the Clinical and Translational Research Unit (CTRU) at the Charlestown Navy Yard campus of MGH.

## What will happen in this research study?

If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures.

Participation in this study will require modifications to your diet during the treatment periods. These modifications also include avoidance of specific foods and drinks throughout your participation. At the start of the study, it is important to:

- Avoid drinking alcohol for 72 hours before all in-person visits.
- Avoid eating grapefruit, pomelo, Seville orange products and drinking Seville orange juices for *14 days* prior to the start of Treatment Period 1.

Further information regarding your diet and foods/drinks you will need to avoid will be covered in detail later in this form.

#### **Screening Period**

#### **Informed Consent Visit (Visit 1a – Virtual)**

The informed consent visit will occur remotely via a secure videoconferencing platform. At this visit you will meet with the Principal Investigator and/or another study investigator to review the study in detail and electronically sign the informed consent form. This virtual meeting will last between an hour to an hour and a half. At this visit the following information will also be collected to start to assess your eligibility to participate in this study:

- Obtain your demographics (statistical data that describes you)
- Review of your medical and surgical history
- Review of your prior medications (taken up to 60 days before signing informed consent) and current medications

#### **Screening Visit (Visit 1b)**

The in-person screening visit will take about 4 hours at the CTRU. At this visit, we will do some tests and procedures to determine if you qualify to take part in this research study. The study




| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

doctor will review the results of these tests and procedures to determine your eligibility to participate in the study. If you do not qualify, the study doctor will tell you why.

At this visit, we will:

- Review the study's Inclusion/Exclusion criteria
- Document any adverse events and review of medications since the virtual Informed Consent visit
- Perform a physical exam (including a brief neurological exam)
- Obtain vital signs (Blood Pressure, pulse rate and body temperature).
- Collect body height and body weight measurements
- Administer mood questionnaires
- Perform an electrocardiogram (ECG)
- Perform a blood draw and collect a urine sample for clinical lab analysis and to test for illicit drugs and alcohol use
- Perform a blood pregnancy test if you are a female and able to become pregnant (Note: Pregnant or breast-feeding females cannot take part in this research study)
- Perform an MRI scan (75 minutes)

These procedures will be scheduled to occur within a one-day study visit, however, in some instances, the screening procedures may be split between two days.

#### **Urine Drug Screening and Alcohol Test**

During this study, we will test your urine for certain illicit drugs (e.g., cocaine, marijuana) and alcohol. If your urine show that you have taken any of these drugs or have consumed alcohol within 72 hours, you cannot be in this study. The results of these urine tests will not become part of your medical record. These test results will, however, remain part of your study record.

#### Electrocardiogram (ECG)

This test checks the electrical activity of your heart. We will place several small, sticky pads on your chest, arms, and legs. Each pad has a wire attached to it. The wires connect to a machine that makes a recording of your heart rhythm. This painless non-invasive test takes about 15 minutes.

#### **Magnetic Resonance Imaging (MRI)**

We will take detailed pictures of your brain using an MRI (magnetic resonance imaging) scan 17 times during this study. During these MRI scans, we will use a specific imaging technique called magnetic resonance spectroscopy (MRS) to explore brain metabolism. An MRI scanner uses a strong magnet and radio waves to take these pictures. Due to this, people who have certain metal implants cannot have this scan. You will be asked to remove all removable metal items (i.e. chains, bracelets, watches, etc.) and clothing before the scan and be given specific pants, shirts, and a robe (if needed) to wear for the procedure.





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

The MRI scanner is a large machine shaped like a tube. You will lie on a narrow table and will be moved into the MRI tunnel. The tunnel is only a little larger than your body. You will be asked to lie still during the scan. Each MRI short scan will take approximately 45 minutes and each MRI long scan will take approximately 75 minutes.

The MRI scanner makes loud banging noises as it takes pictures. We will give you earplugs to reduce the noise. You will be able to hear and speak to the research staff at all times during the scan. We can stop the scan at any time, if needed. You will be given a button while you are in the MRI scanner that you can use to alert the staff if you need to stop or if you are experiencing problems during the scan.

#### **Blood Draws**

We will draw blood from a vein in your arm for standard laboratory tests and to determine how your body uses the study drug at various timepoints throughout the study. Blood will be drawn for safety checks at your screening and follow-up visits. Additional blood will be collected at select study visits to measure levels of study drug in your blood. If any problems arise that are thought to be associated with AL001 and/or Lithium Carbonate, you may have more blood drawn, based on assessment from a study investigator.

#### Breakdown of Blood Draw Amounts

At the Screening visit, we will draw up to 38 mL (about 2.5 tablespoons) of blood from a vein in your arm for clinical safety labs.

Safety labs blood draws occurring at the beginning and at the end of each treatment period will involve drawing up to the following amount of blood, in total:

- Treatment Period 1: up to 19 mL (about 1 1/3 tablespoons)
- Treatment Period 2: up to 24 mL (about 1 2/3 tablespoons)

During each treatment period, there will be 31 blood draws to assess for the presence of the study drugs in your blood. When you are taking AL001, we will draw up to 310 mL (about 21 tablespoons) of blood throughout this treatment period. When you are taking Lithium Carbonate, we will draw up to 190 mL (about 13 tablespoons) of blood throughout this treatment period. Twenty-nine (29) of these draws in each treatment period will occur over a 24-hour period. For these blood draws we will use a blood sparing intravenous catheter for your comfort.

At the in-clinic follow-up visit after Treatment Period 2, we will draw up to 22 mL (about 1 1/2 tablespoons) of blood for clinical safety labs.

In total, up to 603 mL (about 41 tablespoons) of blood will be collected over the course of the entire research study lasting about 4 and a half months.





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

Please note that if you stop participation early, we will perform a blood draw for safety analysis at the Early Termination visit. At this visit, up to 32 mL (about 2 tablespoons) of blood will be drawn from a vein in your arm.

#### **Study Drug Assignment Schedule**

If you qualify for the study, we will assign you by chance (like a coin toss) to start the study in either the AL001 group or the Lithium Carbonate group. You and the study doctor cannot choose your initial study group. You will receive the alternate treatment during the second treatment period. Therefore, you will take both study drugs during the study with an outpatient washout period in between treatments.

#### **Treatment Period 1 (16 days)**

After it is determined that you qualify for the study, you will be scheduled to report to the Translational and Clinical Research Center (TCRC) at the main campus of MGH. You must be admitted by 4pm the day before your first scheduled treatment dose. You will spend 15 days and 14 nights within the TCRC. On the morning of the 15<sup>th</sup> day, you will be transferred to the Clinical and Translational Research Unit (CTRU) at the Charlestown Navy Yard campus of MGH for the last overnight stay.

You will be randomly assigned to take either AL001 or Lithium Carbonate for the entirety of this treatment period. During this treatment period, we will perform specific procedures on the following days:

TCRC Check-in Day (Visit 2; Visit 18 for Treatment Period 2)

- Obtain vital signs
- Document any adverse events and review current medications and medications taken since the last visit
- Collect body weight measurements
- Review the study's Inclusion/Exclusion criteria to confirm continued eligibility to participate in the study
- Perform a blood draw and collect a urine sample for clinical lab analysis and to test for illicit drugs and alcohol use
- Perform urine pregnancy test (if you are a female and able to become pregnant)
- Administer mood questionnaires
- Administer a health status questionnaire
- Once continued eligibility is confirmed, assign a study drug for this treatment period based on the randomization schedule
- Provide a standardized meal (dinner)





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

Treatment Day 1 (Visit 3; Visit 19 for Treatment Period 2)

- Prior to first 8AM dose:
  - Obtain vital signs
  - o Document any adverse events and review of medications taken in the last 24 hours
  - o Perform an ECG
  - o Perform a blood draw for research lab analysis
- Administer three treatments (8AM, 2PM, 8PM) while fasting of either AL001 or Lithium Carbonate capsules
- Provide standardized meals (breakfast, lunch, and dinner)
- After third dose (8PM)
  - Perform an ECG

*Treatment Days 2-12 (Visits 4 to 14; Visits 20 to 30 for Treatment Period 2)* 

- Prior to first 8AM dose:
  - Obtain vital signs
  - o Document any adverse events and review of medications taken in the last 24 hours
- Administer three daily treatments (8AM, 2PM, 8PM) while fasting of AL001 or Lithium Carbonate capsules
- Administer a mood questionnaire (this will occur on *at least* two separate days during the treatment period)
- Provide standardized daily meals (breakfast, lunch, and dinner)

Treatment Day 13 (Visit 15; Visit 31 for Treatment Period 2)

- Prior to first 8AM dose:
  - Obtain vital signs
  - o Document any adverse events and review of medications taken in the last 24 hours
  - o Perform an ECG
  - o Perform a blood draw for research lab analysis
- Administer three treatments (8AM, 2PM, 8PM) while fasting of AL001 or Lithium Carbonate capsules
- Provide standardized meals (breakfast, lunch, and dinner)

Treatment Day 14 (Visit 16; Visit 32 for Treatment Period 2)

- Transfer from TCRC (MGH Main Campus) to CTRU in Charlestown
- Prior to first 8AM dose:





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

- Obtain vital signs
- o Document any adverse events and review of medications taken in the last 24 hours
- o Perform an ECG
- o Perform a blood draw for research lab analysis
- o Perform an MRI scan within 1 hour before 1st dose of the day (45 mins)
- Administer three treatments (8AM, 2PM, 8PM) while fasting of either AL001 or Lithium Carbonate capsules
- Perform repeated blood draws (28 total) over the next 24 hours after first 8AM dose
- Perform repeated MRI scans (7 total) over the next 24 hours after first 8AM dose (one scan will be about 75 minutes and the other 6 scans will be about 45 minutes each)
- Provide standardized meals (breakfast, lunch, and dinner)
- Overnight Stay at CTRU

#### Day 15 (Visit 17; Visit 33 for Treatment Period 2)

- No treatment will be administered on this day
- Obtain vital signs
- Document any adverse events and review of medications taken in the last 24 hours
- Perform an ECG
- Perform a physical exam (including a brief neurological exam)
- Collect body weight measurements
- Perform a blood draw for clinical and research lab analyses
- Collect a urine sample for clinical lab analysis
- Administer mood questionnaires
- Provide a standardized meal (breakfast)
- Discharged from the clinic

Please note: The 5<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> MRIs as well as the 20<sup>th</sup> through 28<sup>th</sup> blood draws will occur overnight into the morning of Day 15 (Visit 17).

#### **Washout Period**

After clinic discharge from Treatment Period 1, you will enter a "Washout Period" where you will no longer be taking the study drug from Treatment Period 1. This washout period will last between 9 to 28 days and will allow the drug from Treatment Period 1 to leave your body before beginning Treatment Period 2. During this time a study staff member will call you twice, at a minimum, to check in. These phone calls will occur about 2-3 days after completing Treatment Period 1, then every 5-7 days until you return to the TCRC (at MGH main campus) for Treatment Period 2; however, the timing of these phone calls may vary. During these calls we will ask you to complete some questionnaires over the phone.





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

#### **Treatment Period 2 (16 days; Visits 18 to 33)**

During Treatment Period 2, you will again be admitted into the TCRC (at MGH main campus) for 15 days and 14 nights (*TCRC Check-In Day* to *Treatment Day 14*). Again, there will also be an overnight stay at the CTRU in Charlestown for the last overnight stay (*Treatment Day 14* to *Day 15*). The same procedures performed during Treatment Period 1 will be performed during this period; however, you will be taking the other study drug. In other words, you will either take AL001 or Lithium Carbonate for the entirety of this period, depending on which drug you took during Treatment Period 1.

On Day 15 of Treatment Period 2 (Visit 33), we will also perform a urine pregnancy test if you are a female and able to become pregnant.

#### **Taking the Study Drug**

You will take each of the study drugs by mouth three times a day with 240 mL of non-carbonated water. All doses will be taken under fasted conditions (i.e., 1 hour before or 4 hours after meals) at 8AM, 2PM, and 8PM (6 hours apart, within  $\pm 10$  minutes). Water will be allowed as desired except for 1 hour before and after drug administration. It is important that you follow our instructions about how to take the study drug. A mouth check will be performed by a study staff after each dose to ensure that you have swallowed all the capsules.

#### General Information about Study Participation and Each Treatment Period

During each treatment period you are allowed to:

- Have visitors (one person at a time)
- Bring items to keep you busy (e.g., crafts, books, laptop, etc.)
- Shower make sure you bring shower shoes and a hair dryer
- Do laundry with the help of a study staff member
- Go on supervised short walks on the campus grounds with a study staff member or an MGH staff member

During each treatment period you are **not** allowed to:

• Leave the TCRC or MGH campus unsupervised

#### **Standardized Meals During Treatment Periods**

During each Treatment Period, your meals will be standardized. This means that each breakfast, lunch, and dinner will be consistent based on your choices starting at your TCRC Check-in Day. You will work with a dietitian to create a meal plan for both of your stays. This meal plan will remain the same throughout each of the 16-day Treatment Periods. Depending on the timing of study drug doses and meals throughout the day, snacks can also be provided at the judgement of the study staff.





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

#### Foods and Drinks to Avoid During your Participation

In addition to your standardized meals during each treatment period, there are specific foods you must avoid throughout your participation in the study, *including during the washout period*.

- Avoid drinking alcohol for at least <u>72 hours</u> before each in-person study visit and during each Treatment Period. In general, during the times where you could consume alcohol, you should avoid drinking more than 2 standard drinks in one sitting.
- Avoid consuming (eating or drinking) Poppy seeds and Quinine (tonic water) within <u>48</u> <u>hours</u> of Treatment Day 1 until the end of your participation in the study, *including during the washout period*.
- Avoid consuming (eating or drinking) caffeine <u>48 hours</u> before your check in day for Treatment Period 1 until your completion of Treatment Period 2. This includes also avoiding caffeine during the washout period. Caffeine can be in coffee, energy drinks, soda, and chocolate, among other foods and drinks.
- Refrain from consuming the following for at least <u>14 days</u> prior to your check in day for Treatment Period 1 until your completion of Treatment Period 2, *including during the washout period*:
  - o Grapefruits
  - o Pomelos
  - Seville Orange products and juices

Please inform a study staff member if you do eat or drink any of the above-mentioned foods or drinks. Please also inform a study staff member if you happen to eat or drink anything outside of your standardized meal plan during your Treatment Periods at the TCRC or during your overnight stays at the CTRU.

#### Follow-Up Period

The follow-up period consists of an in-person visit to the CTRU in Charlestown and a telephone call.

*In-Clinic Follow-up Visit (Visit 34)* 

This visit will take place approximately 7 days after completion of Treatment Period 2. This visit will last up to 2 hours and involve the following procedures:

• Obtain vital signs




| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

- Document any adverse events and review of medications since the last visit
- Perform an ECG
- Perform a physical exam (including a brief neurological exam)
- Collect body weight measurements
- Perform a blood draw and collect a urine sample for clinical lab analysis
- Perform a urine pregnancy test (if you are a female and able to become pregnant)
- Administer mood questionnaires
- Administer a health status questionnaire

#### Telephone Follow-up Call (Visit 35)

This phone call will occur approximately 27 days after completion of Treatment Period 2. This will serve as your last day of study participation. This phone call will last about 30 minutes and include the following procedures:

- Document any adverse events and review of medications since the last visit
- Administer a mood questionnaire
- Administer a health status questionnaire

If any lab results from the blood draw performed at the in-clinic follow-up visit (Visit 34) are found to be clinically significant with reasonable possibility for this clinical finding to be caused by the study drug, then we will ask you to come in person for a repeat blood draw. This significant finding will be followed until resolved.

#### **COVID-19 Testing (if applicable)**

At the discretion of the investigator, you may undergo testing for COVID-19 throughout the study. This will be based on local health policies and guidance at the time of your participation and if there is any suspected or known contact with an individual infected with COVID-19. The same principles apply to testing for other emergent infectious diseases and illnesses.

#### **Early Termination (if applicable)**

An in-person Early Termination Visit will take place if you decide to stop taking part in the study for any reason after starting treatment, but prior to completing all study procedures. This visit will take approximately 1 ½ hours at the CTRU in Charlestown and involve the following procedures:

- Obtain your vital signs
- Document any adverse events and review of medications since the last visit
- Perform a physical exam (including a brief neurological exam)
- Collect body weight measurements
- Perform an ECG
- Perform a blood draw and collect a urine sample for clinical and research lab analyses
- Perform a urine pregnancy test (if you are a female and able to become pregnant)




| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

- Administer mood questionnaires
- Administer a health status questionnaire

Also, the study doctor may take you out of the study without your permission. This may happen because:

- The study doctor thinks it is best for you to stop taking the study drug
- You cannot make the required study visits
- You failed to continue to meet the study eligibility criteria
- You were non-compliant or violated protocol restrictions
- The sponsor decides to stop the study
- We stop conducting the study for other reasons

If this happens, the study doctor will explain why you need to stop taking part in the study. We will ask you to come in for a final study visit as described above.

## Review of Medical Records from Hospital Admissions or Emergency Department Visits

Mass General Brigham has an electronic system that lets your study doctors know if you are admitted to a Mass General Brigham Hospital, or if you visit a Mass General Brigham Hospital Emergency Department. We want to make sure the study doctors know about any possible problems or side effects that you experience while you are taking part in the study.

## Study Information Included in Your Electronic Medical Record

A notation that you are taking part in this research study may be made in your electronic medical record. Information from the research that relates to your general medical care may be included in the record (for example: list of allergies, results of standard blood tests done at the hospital labs).

Please ask your study doctor if you have any questions about what information will be included in your electronic medical record.

## Sending Study Information to Research Collaborators Outside Mass General Brigham

We will label all your study materials with a code instead of your name. The key to the code connects your name to your study information and samples. We will keep the key to the code here at Mass General Brigham and will not share it with our research collaborators. No one outside of Mass General Brigham will know which study information or samples are yours.

We will securely send your study information and/or samples to Alzamend Neuro, Inc. All information sent to Alzamend Neuro, Inc. will not include any private health information (PHI).





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

Laboratory samples will sometimes be sent to outside laboratories for analysis. However, these samples will not contain your name or identifying information. This study will also have a safety monitor, or someone not performing the research who oversees the data and safety of participants. This medical monitor will see all study data, some of which may include PHI such as date of birth, medical record number (MRN) and name as this information is needed for some study visit documents.

## How may we use and share your samples and health information for other research?

The samples and information we collect in this study may help advance other research. If you join this study, we may remove all information that identifies you (for example your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It will not be possible to link the information or samples back to you. Information and/or samples may be shared with investigators at our hospitals, at other academic institutions or at for-profit, commercial entities. You will not be asked to provide additional informed consent for these uses.

### Will you get the results of this research study?

No. The research study we are doing is only a steppingstone in understanding the safety and effects of AL001 when compared to Lithium Carbonate. Therefore, no information about the results of this research study or the results of your individual participation in the research study will be given to you or your doctor. Tests done for the research using your samples will not be useful in directing your medical treatment. The results of the tests will not be placed in your medical record.

# What are the risks and possible discomforts from being in this research study?

### **Risks of Taking AL001**

AL001 is composed of Lithium and Salicylate, and an amino-acid, L-proline, that is an essentially needed dietary component commonly found in foods. Taking AL001 may cause you to have one or more of the side effects listed below.

Common side effects of Lithium:

- Headache
- Mild to moderate nausea or vomiting
- Diarrhea
- Dizziness
- Drowsiness
- Changes in appetite
- Hand tremors




General Template - Drug Clinical Trial

**Version Date: November 2022** 

| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

- Dry mouth
- Increased thirst
- Increased urination
- Hair thinning/hair loss
- Acne-like rash

#### Less common side effects of Lithium:

- Severe nausea and vomiting
- Severe hand tremors
- Confusion
- Vision changes
- Unsteadiness while walking

#### Uncommon side effects of Lithium:

Diabetes

#### Common side effects of Salicylate:

- Indigestion
- Ringing in the ears
- Heartburn
- Nausea

#### Less common side effects of Salicylate:

- Mild to moderate vomiting
- Anorexia
- Abdominal pain

There may be other risks of AL001 that are currently unknown.

#### **Risks of Taking Lithium Carbonate**

Taking Lithium Carbonate may cause you to have one or more of the side effects listed below.

#### Common side effects of Lithium Carbonate:

- Muscle tremors or twitching, usually in the hands
- Dizziness
- Drowsiness
- Trouble walking
- Increased urination




| Subject | Name: | |
|---------|-------|------------------------|
| MRN or | DOB: | |
| | | Subject Identification |

- Increased thirst, dry mouth
- Nausea, vomiting
- Appetite changes
- Rash
- Blurred vision

#### Less Common side effects of Lithium Carbonate:

- Headache
- Diarrhea
- Abdominal pain
- Dry or thinning hair
- Confusion, poor memory
- Fainting
- Irregular heartbeat
- Stiffness in the arms or legs
- Trouble breathing particularly with physical exercise
- Weight gain or loss
- Indigestion
- Cough
- Fever
- Agitation
- Swelling of the ankles or wrists

#### Rare Side effects of Lithium Carbonate:

- Blue color and pain in fingers and toes
- Eye pain
- Ringing in the ears

As with any drug, an allergic reaction can occur. Allergic reactions can be mild or more serious, and can even result in death. Common symptoms of an allergic reaction are rash, itching, skin problems, swelling of the face and throat, or trouble breathing. If you think you are having an allergic reaction, alert the study doctor and or study staff right away. If you are having trouble breathing, call 911 immediately.

#### Risks of Taking Other Medications with either AL001 or Lithium Carbonate





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

Various drug types have been known to have significant interactions with lithium.

For your safety during this study, call your study doctor **BEFORE** you take any:

- new medications prescribed by your own doctor
- other medications sold over-the-counter without a prescription
- dietary or herbal supplements

Please note that if you do start taking a new medication either prescribed or over the counter while you are participating in this study, even in the washout period, you may be unable to continue your participation. Please inform the study doctor or a staff member if you may be starting any new medication while participating in the study.

Only a small number of people have taken AL001. Therefore, we don't know about all the side effects that can happen when taking AL001 with other drugs. Due to this and the fact that other products may affect AL001 and Lithium Carbonate, we kindly ask that you refrain from taking, eating, or ingesting any of the following products:

| Product | Restriction Time Before<br>Treatment Period | Restriction Time During Treatment and Participation |
|---|---|---|
| Prescription Drugs and St. | 14 days prior to TCRC | Throughout study |
| John's Wort | Check-in Day | participation, including |
| | | during the washout period |
| Over the counter (OTC) drugs, including cold preparations, acetaminophen (for example, Tylenol), anti-inflammatory drugs (for example, Advil, Motrin), vitamins, and natural products used for therapeutic benefits, and antacid preparations | 14 days prior to the in-person<br>screening visit and 14 days<br>prior to TCRC Check-in Day | Throughout study participation, including during the washout period |
| Salicylate-containing product (for example, Aspirin) other | 7 days prior to first study | Throughout the study (including during the washout |
| than low dose aspirin for cardio (heart) protection | drug dose (Treatment Day 1) | period) until 7 days after the last study drug administration |
| Alcohol-based products | 72 hours before study visits | Throughout study participation |





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

| Product | Restriction Time Before<br>Treatment Period | Restriction Time During Treatment and Participation |
|---|---|---|
| Products containing caffeine/xanthines (for example, coffee, tea, chocolate, cola, caffeine-containing soda like Mountain Dew, Dr. Pepper, beverages and energy drinks such as Red Bull, Extreme Energy Shot and Guru) | 48 hours prior to TCRC<br>Check-in Day | Throughout study participation, including during the washout period |
| Products containing poppy seeds or quinine (tonic water) | 48 hours prior to the first study drug dose (Treatment Day 1) | Throughout study participation, including during the washout period |
| Products containing pomelo,<br>grapefruit and/or Seville<br>orange products, or juice | 14 days prior to TCRC<br>Check-in Day | Throughout study participation, including during the washout period |

#### **Risks of Blood Draws**

You may have a bruise (a black and blue mark) or pain where we take the blood samples. There is also a small risk of infection, lightheadedness, and/or fainting.

#### Risks of Magnetic Resonance Imaging (MRI)

MRIs uses powerful magnets to make images. There are no known radiation risks associated with MRI. However, people with metal implants such as surgical clips or pacemakers should not have MRIs. All credit cards and other items with magnetic strips should also be kept out of the MRI room. People who feel uncomfortable in confined spaces (claustrophobia) may feel uncomfortable in the narrow tube. The MRI makes loud banging noises as it takes images. Earplugs will be used to reduce this noise. The MRI can be stopped at any time at your request. You will be given a button you can press at any time to talk to the MRI and study staff.

If you are or suspect you are pregnant, you should not participate in this study. The MRI has the potential during routine use to cause localized warming of your skin and underlying tissues. You should immediately inform us if you experience discomfort due to warming and the procedure will be stopped.

Some people may experience dizziness or rarely nausea when going into an MRI scanner and these sensations may be more common in scans with higher magnetic fields. In most cases, these symptoms only last a short time. However, some people may experience them throughout the scan





| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

and/or continue to experience them for a short period of time after; generally, less than half an hour. No case of permanent problems is known.

Scanning may take up to 75 minutes. You will be required to lie still for much of this time. Some people may find it uncomfortable lying still for such long periods of time. Others may feel uncomfortable with the narrow dimensions of the scanner or find the loud scanner noises unpleasant. If you feel uncomfortable, you may request that scanning be stopped at any time.

#### **Risk of Overnight Hospital Stay**

You may become frustrated or experience feelings of isolation or loneliness during the extended overnight stays at the TCRC. Please talk to a study staff member or a member of the TCRC if these feelings become intense or unmanageable.

#### **Risks of Questionnaires**

Questionnaires may cause you to feel sad or upset. Study personnel are experienced with such evaluations and sensitive to these issues; also you are free to cease or take a break from the questionnaire sessions at any time.

#### **Data Security Risks**

Study data that we collect throughout your participation in the study will be stored within QMENTA Imaging Hub and REDCap Cloud. These are secured database platforms and only necessary study staff and qualified QMENTA and REDCap personnel will have access to data collected within this study. Your study data will be identified within the study database by using a unique study ID. Your name, date of birth, and general contact information (e.g., email, telephone number, address) will be collected and stored within the study database, however, no other personal identifiers will be collected. The risk is very small; however, data security breaches are always a risk when using electronic based systems. Every precaution will be put in place by QMENTA, REDCap, and the MGH staff to ensure your privacy and confidentiality are protected both during and after your study participation. Any data shared with the sponsor or laboratories used for blood specimen processing will only contain your unique study ID and no identifiable information.

## Safety Procedures for Female Participants Who are Able to Become Pregnant

If you are a menopausal woman and have not had a menstrual period for the past 12 months or more, you will not need to have a pregnancy test. Also, if you have had any well-documented method of surgical sterilization, you will not need to have a pregnancy test. Methods of surgical sterilization include having had a hysterectomy (removal of the uterus), bilateral oophorectomy (removal of both ovaries), a tubal ligation (having your tubes tied), and transvaginal occlusion (plugging the opening of the tubes with a coil). All other female subjects must have a negative pregnancy test before starting the study drug.




| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

If you are sexually active and able to become pregnant, you must agree to use one of the birth control methods listed below. You must use birth control starting at the screening visit until 30 days after your last dose of study drug in Treatment Period 2.

Acceptable birth control methods for use in this study are:

- hormonal methods, such as birth control pills, patches, injections, vaginal rings, or implants
- barrier methods (such as a condom, cervical cap, or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- intrauterine device (IUD)
- abstinence (no sex)

If you miss a period, or think you might be pregnant during the study, you must tell the study doctor immediately. If you become pregnant, you must stop taking the study drug and stop taking part in the study. The study doctor may ask for your permission to collect information about the outcome of your pregnancy and the condition of your newborn.

#### Safety Procedures for Male Participants Who are Able to Father a Child

If you are sexually active and able to father a child, you must agree to use one of the birth control methods listed below. You must use birth control starting at the screening visit until 30 days after your last dose of the study drug in Treatment Period 2.

Acceptable birth control methods that you can use in this study are:

- condoms with spermicide (a foam, cream, or gel that kills sperm)
- abstinence (no sex)

Acceptable birth control methods that your partner(s) should use are:

- hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- barrier methods (such as a condom, cervical cap, or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- intrauterine device (IUD)

If your female partner becomes pregnant during your participation in the study or within 90 days of study completion, the sponsor, Alzamend Neuro, Inc., would like to follow the outcome of the pregnancy. You should notify us immediately if your partner becomes pregnant. We will work with you and your female partner to provide contact information to the sponsor. She may be asked to sign a release of medical information form that gives her doctors permission to provide information to the sponsor. You will not have to stop taking the study drug or stop taking part in the study if your partner becomes pregnant.

## What are the possible benefits from being in this research study?





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

You will not benefit from taking part in this research study. However, others with psychiatric and neurological conditions may benefit in the future from what we learn in this study.

## Can you still get medical care within Mass General Brigham if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Mass General Brigham now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

#### What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop your participation in the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?

We will pay you up to \$10,300 if you complete the study. You will be paid after completion of Baseline MRI scan, Treatment Period 1, Treatment Period 2, and then again after completion of the full study. If you do not complete the study, we will prorate your compensation for all the visits and or procedures you completed. Compensation breakdown for specific procedures is as follows:

- Baseline MRI scan \$100
- Treatment Period 1
  - o TCRC Overnight Stays \$200/day (\$2800 total)
  - o CTRU Procedures on Day 14 & Day 15 \$800
    - Repeated PK Blood Draws (29): \$25/draw (\$725 total)
    - Day 15 CTRU Procedures: \$75
  - o 7 Short MRI scans \$700 (\$100 for each completed scan)
  - o Long MRI scan \$100
  - o Total for Treatment Period 1: \$4,400
- Treatment Period 2
  - o TCRC Overnight Stays \$200/day (\$2800 Total)
  - CTRU Procedures on Day 14 & Day 15 \$800





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

- Repeated PK Blood Draws (29): \$25/draw (\$725 total)
- Day 15 CTRU Procedures: \$75
- o 7 Short MRI scans \$700 (\$100 for each completed scan)
- o Long MRI scan \$100
- o Total for Treatment Period 2: \$4,400
- Completion Bonus: \$1,400
  - Note: You will only receive the completion bonus if and only if you complete all other procedures in the study. This includes Treatment Period 1, the Washout Period, Treatment Period 2, and the Follow-up visits in full. No exceptions will be made.

We will pay for transportation to and from the hospital for the drug treatment periods. If you are coming from out of state or live over 2 hours away by car, you will be given the option to stay overnight in a hotel before traveling home after each treatment period.

We will also reimburse you up to \$50 for any laundry you do during the Treatment Periods.

We may use your samples and information to develop a new product or medical test to be sold. The sponsor, hospital, and researchers may benefit if this happens. There are no plans to pay you if your samples are used for this purpose.

## What will you have to pay for if you take part in this research study?

Alzamend Neuro, Inc. is providing the study drugs at no cost.

Study funds will pay for study-related procedures and study visits that are done only for research.

Study funds will pay for certain study-related items and services. We may bill your health insurer for, among other things, routine items and services you would have received even if you did not take part in the research. You will be responsible for payment of any deductibles and co-payments required by your insurer for this routine care or other billed care. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in Patient Financial Services about these costs.

## What happens if you are injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

In this study, Alzamend Neuro, Inc. will pay for medical treatment for any injury that is not paid for by your health insurer if the injury is a direct result of your taking part in the study. Alzamend Neuro, Inc. has no plans to offer you any other payments or other type of compensation.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

## If you take part in this research study, how will we protect your privacy?

Federal law requires Mass General Brigham to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information".

#### In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

## Who may see, use, and share your identifiable information and why they may need to do so:

- Mass General Brigham researchers and staff involved in this study
- The sponsor(s) of this study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Mass General Brigham ethics board or an ethics board outside Mass General Brigham that oversees this research
- A group that oversees the data (study information) and safety of the study
- Non-research staff within Mass General Brigham who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)
- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of





| Subject Name: |
|------------------------|
| MRN or DOB: |
| Subject Identification |

Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records

• Public health and safety authorities, if we learn information that could mean harm to you or others (such as to make required reports about communicable diseases or about child or elder abuse)

• Other: N/A

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your identifiable information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your identifiable information for any mailing or marketing list. However, once your information is shared outside Mass General Brigham, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your health information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifying information **will not** be used for these purposes without your specific permission.

#### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your health information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your health information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.





| C. L. AN | |
|---------------|------------------------|
| Subject Name: | |
| MRN or DOB: | |
| | Subject Identification |
| | Subject Identification |

You have the right to see and get a copy of your health information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.




| Subject Name: | |
|---------------|------------------------|
| MRN or DOB: | |
| | Subject Identification |

#### **Informed Consent and Authorization**

#### **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

## Signature of Subject:

| | | Signature of Subject. |
|---|---|---|
| I give my consent to take part in this research study and agree to allow my health information be used and shared as described above. | | |
| Print Name of Subject | | |
| Subject Signature | <br>Date | Time (optional) |
| Signature of Study Doctor or Pe | rson Obtaining Cons | ent: |
| Statement of Study Doctor or Person | <b>Obtaining Consent</b> | |
| <ul> <li>I have explained the research to</li> </ul> | | |
| <ul> <li>I have answered all questions about</li> </ul> | out this research study to t | he best of my ability. |
| I have answered all questions about Print Name | out this research study to t | he best of my ability. |


IRB Protocol No: 2024P003031 IRB Expiration Date: 3/5/2026
Consent Form Valid Date: 5/21/2025 IRB Submission: AME4

Consent Form Version: April 21st, 2025